CLINICAL TRIAL: NCT04494204
Title: An Open Label, Multicenter, Randomized, Controlled, Clinical Study to Evaluate the Efficacy and Safety of a Combination of Treatment of Reginmune Capsule and Immunofree Tablets Compared With Standard Treatment Protocol in the Treatment of Mild to Moderate COVID-19 Patients.
Brief Title: Effect of a Combination of Treatment of Reginmune Capsule and Immunofree Tablets in the Treatment of Mild to Moderate COVID-19 Patients
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: PUNEET MITTAL (Network)
Responsible Party: Sponsor-Investigator, PUNEET MITTAL, Clinical Research Consultant, Nutrin GmbH
Organization: Nutrin GmbH (Network)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MGCTS/20/105
Record Dates: First submitted 2020-07-28; First posted 2020-07-31 (Actual); Last update posted 2020-12-22 (Actual); Status verified 2020-12

CONDITIONS: Treatment of Covid-19 Virus Infection
Keywords: coronavirus; covid-19; covid; corona; coagulation; immunofree; mgcts; biogetica
MeSH Terms: conditions — Coronavirus Infections; COVID-19; Thrombosis

STUDY DESIGN:
Intervention Model Description: After obtaining the informed consent, patients will be screened by undergoing various assessments and after confirming eligibility, eligible patients will be randomized in the study and assigned either to the test group or control group with Best standard of care as per institutional practice, for 10 days treatment period. Patient will be hospitalized during the treatment period.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): 2 tablets Immunofree 500 mg tablets thrice a day for 10 days and 1 capsule Reginmune 750 mg twice a day for 10 days
  Interventions: Combination Product: Immunofree tablets and Reginmune capsule
- Comparator Agent (Active Comparator): As per standard National Clinical Management Protocol for COVID-19 by Government of India, Ministry of Health and Family Welfare, Directorate General of Health Services, (EMR Division), Version 3, 13.06.20
  Interventions: Combination Product: Immunofree tablets and Reginmune capsule

INTERVENTIONS:
Combination Product: Immunofree tablets and Reginmune capsule — 2 Immunofree tablets thrice a day at an interval of 4-5 hours for 10 days and 1 Reginmune capsule twice a day for 10 days

SUMMARY:
While novel drug discovery and vaccine studies are time taking process, re-purposing old drugs against the COVID-2019 epidemic can help identify treatments, with known pre-clinical, pharmacokinetic, pharmacodynamic, and toxicity profiles, which can rapidly enter Phase 3 or 4 or can be used directly in clinical settings. Immunofree has many of the herbs which have been evaluated by other trials published for Covid-19 treatment.

The Immunofree tablet of the test product is an Ayurvedic proprietary medicine and is a combination of polyherbal mixture. The components of this formulation are known for their anti-viral and immunomodulatory effects. Also, Reginmune, owing to its immunomodulatory effect might help in easing the symptoms and decrease the viral load.

DETAILED DESCRIPTION:
The symptoms of COVID-19 are mainly for respiratory disorders and similar to severe acute respiratory symptoms. The common signs of infection observed in COVID-19 patients include respiratory symptoms, sneezing, fever, cough, shortness of breath and other breathing difficulties. In case of severely infected patients, infection can cause pneumonia, severe acute respiratory syndrome (SARS), kidney failure and even death in many cases. There are many people who had high viral load but do not develop COVID-19 symptoms like coughing or sneezing. Such asymptomatic people serve as hidden carriers of virus and may further contribute in enhanced transmission of virus to other people. In absence of any emergency medicine or complete therapy for COVID-19; the prevention of spread of SARS-CoV2 virus and regulation of infection is the prime step in controlling this epidemic disease, in which the test products can be of immense value.

The test product, Capsule Reginmune is a combination of some phytochemicals, amino acids, vitamins and minerals and a bio-polymer in cellular matrix. The components and their pharmacological activities are as follow:

Echinacea is one of the more popular herbal supplements suggested for boosting immunity. Some respiratory and antiviral research has also been done on Echinacea. Echinacea is not mentioned by the Indian and Chinese Governments however in their guidelines for boosting immunity.

Cats Claw (Uncaria Tomentosa)has shown potent anti-viral and immunomodulatory activity in a recent study. The results demonstrated an in vitro inhibitory activity by both extract and alkaloidal fraction, reducing DENV-Ag+ cell rates in treated monocytes. A multiple microbead immunoassay was applied for cytokine determination (TNF-alpha, IFN-alpha, IL-6 and IL-10) in infected monocyte culture supernatants. The alkaloidal fraction induced a strong immunomodulation: TNF-alpha and IFN-alpha levels were significantly decreased and there was a tendency towards IL-10 modulation. The researchers conclude that the alkaloidal fraction was the most effective in reducing monocyte infection rates and cytokine levels. The antiviral and immunomodulating in vitro effects from U. tomentosa pentacyclic oxindole alkaloids displayed novel properties regarding therapeutic procedures in Dengue Fever and might be further investigated as a promising candidate for clinical application.

Vitamin C: Well accepted to increase immunity and an effective antiviral. However, not many people realize the vast difference in food derived vitamin C and ascorbic acid which is a dead synthesized molecule used to clean pools. Therefore, it is strongly recommended that one should only take food derived Vitamin C.

Zinc: There is some evidence suggesting Zinc can shorten duration of the common cold and one study done in 2010 showing that Zinc had an effect on the older versions of Corona virus. An abundance of evidence has accumulated over the past 50 years to demonstrate the antiviral activity of zinc against a variety of viruses, and via numerous mechanisms. Clinical trial data support the value of zinc in reducing the duration and severity of symptoms of the common cold when administered within 24 hours of the onset of common cold symptoms. However, one must be careful as not all zinc is equally bioavailable and more than 150 mg of Zinc can lead to toxicity.

Copper: A study suggested that copper deficiency may lead to reduction in the number of T cell lymphocytes and impaired host defense against infectious organisms.

L- Lysine: Studies shows L-Lysine supplements may help to boost immunity against certain viral infections.

Aloe Vera: Numerous studies for influenza and herpes has shown that Aloe polysaccharides (APS) extracted from Aloe vera leaves have evident effects on the therapy of virus infection.

Lglutamine: Glutamine is the most abundant and versatile amino acid in the body. Glutamine is currently part of clinical nutritional supplementation protocols and/or recommended for immune suppressed individuals.

L Arginine: Studies have shown that arginine suppressed the growth of HSV-1, concentration dependently and it can boost the activity of T-cells.

L Isoleucine : It has shown to be effective against rotavirus infection. Magnesium Gluconate: It has shown some immunomodulatory effects which was measured by Natural Killer cells activities and phagocytosis.

Sodium Hyaluronate: Hyaluronic acid (HA), one of the main components of extra-cellular matrix and most notably of the fundamental substance of conjunctive tissues, is not an inert structure. Conversely, it displays important biological properties and plays a significant role in crucial physiological processes especially when cellular plasticity is involved such as inflammation, immune reactions, angiogenesis and would healing. It is also strongly involved in neoplastic cells migration and therefore in metastatic spreading of malignant tumors.

The Immunofree tablet of the test product is an Ayurvedic proprietary medicine and is a combination of polyherbal mixture. The components of this formulation are known for their anti-viral and immunomodulatory effects.

Kalmegh also known as Andrographis paniculata has been used in Ayurveda and other herbal traditions for boosting up the immune system. It is believed that the herb has potential antiviral and immunomodulatory properties owing to it containing andrographolide. The following studies are done on it which suggest potential benefit.

Bhumyamalaki: It is also known as Phyllanthus niruri. It seems to exhibit anti-viral anti-inflammatory activity. The following studies for SARS suggest that this may be of benefit.

Glycyrrhiza glabra is also known as licorice, mulethi, etc. It has been used in TCM, Ayurveda and other herbal traditions for lung health and stomach health. It is very alkalizing. It is believed that it has strong antiviral properties and hence this herb is in both Chinese and Indian recommendations. This herb contains glycyrrhizin which showed remarkable qualities in SARS research.

Some reports suggest that strong extracts of this herb are central to the Chinese strategy in Wuhan. The following studies are done on it, which suggest potential benefit.

Tulsi is also known as Ocimum sanctum has been used traditionally in India. It is considered a sacred herb in Ayurveda.Following studies are done on it which suggest potential benefit.

Giloy is also known as Tinospora cordifolia has been used traditionally in Ayurveda as it helps in boosting gut immunity.

Pushkarmool: It is also known as Inula racemosa and it may be an effective herb for flu symptoms. It also supports the normal functioning of the respiratory system.

The drug Pushkarmool has been used in the indigenous system of medicine for a long time. Pushkarmool has been reported in the texts of Ayurveda as possessing Tikta, Katu and Ushna Virya and beneficial for the diseases of heart, throat. It is known to act as an expectorant. It is also used in Ayurveda as an expectorant and resolvent in indurations. Its pharmacological activities include cardioprotective activity, antiallergic activity, antimutagenic and antiapoptotic effects, anti-inflammatory & analgesic effect, adrenergic beta blocking activity.

Alpinia galanga is also known as rasna, sugandhimool, etc. It has been used inTCM, Ayurveda and other herbal traditions for lung health and the potential to reduce the inflammatory process. It is believed that the herb has antiviral activity in human respiratory syncytial viruses. The following studies are done on it which suggest potential benefit.

Draksha: It is also known as Vitis Vinifera. Studies suggeset that the herb possesses a broad spectrum of pharmacological and therapeutic effects such as antioxidative, anti-inflammatory, and antimicrobial activities.

Haldi is also known as Turmeric, Curcuma longa, etc. Alkaloids derived from turmeric have shown potentially strong inhibitory effects on the neuraminidases from two influenza viral strains. The following studies are done on it which suggest potential benefit.

Haritaki is also known as Terminalia chebula has been used in TCM, Ayurveda, and other herbal traditions for boosting immunity. The herb is also possibly useful for easing the symptoms associated with respiratory illnesses. The following studies are done on it which suggest potential benefit.

Aloe Vera: Studies show that extracts of Aloe Vera may help to inhibit the activity of the virus and support the functioning of the lungs.

Shilajit: It is also known as Asphaltum: It has been used traditionally by the Indian Ayurvedic and Siddha systems of traditional medicine to enhance the quality of life. Studies show that the minerals in Shilajit may also possesses immune boosting activities.

Pippali: It is also known as Piper longum. It has been used traditionally in the Ayurvedic system for lung health. Studies suggest that it may help to improve lung function.

Shaival: It is also known as Asthaxantin. Studies show that it may possess antimicrobial and anti-inflammatory properties.

Damanaka - Also known as Artemisia, has potential anti-malarial properties.

ELIGIBILITY:
Inclusion Criteria:

* Gender: Either male or non-pregnant, non-lactating female aged > 18-70
* Patients with RT-PCR confirmed diagnosis of COVID-19
* Patients with mild to moderate COVID-19 infection having either one of the following criteria: oPaO2/FiO2:200-300 OR Respiratory rate ? 24/min and SaO2/SpO2 > 90% on room air
* Subjects willing to give written informed consent
* Subjects able to take the drug orally and comply with the study protocol
* Women of child bearing potential must have a negative urine pregnancy test prior to study entry

Exclusion Criteria:

* Patients with persistent vomiting
* Critically ill patients
* P/F ratio less than 200 (moderate-severe ARDS)
* Shock (Requiring Vasopressor to maintain a MAP more than 65 mm of hg or MAP below 65)
* Patients with known active hepatitis, tuberculosis and definite bacterial or fungal infections
* Patients with altered mental state
* Patients with multiple organ failure requiring ICU monitoring and treatment
* Patients with respiratory failure and requiring mechanical ventilation
* Patients with any concurrent medical condition or uncontrolled, clinically significant systemic disease (e.g. heart failure, hypertension, liver disease, diabetes, anemia etc.) that, in the opinion of investigator precludes the subject's participation in the study or interferes with the interpretation of the study results.
* Patients with history of serology tests positive for hepatitis B, hepatitis C, or human immunodeficiency virus.
* Patients who have received specific antiviral drugs ritonavir/lopinavir, or chloroquine, hydroxychloroquine, azithromycin, monoclonal antibodies within 1 week before admission
* Patient who have participated in another investigational study within 3 months prior to enrollment in this study
* Investigators, study personnel, sponsor's representatives and their first-degree relatives.
* Pregnant subjects

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-08-07 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-20 (Actual)

PRIMARY OUTCOMES:
Time (Days) to clinical improvement from study enrollment | Day 0 - Day 10
  This includes overall time it takes for negative covid-19 results, improvement based on a customized questionnaire for fever, cough, body ache, loss of taste or smell, or other similar conditions

SECONDARY OUTCOMES:
Proportion of participants in each group with oxygen saturation more than 94% on room air for more than 24h | Day 0, Day 5±1 and Day of discharge i.e Day 10±1
  Being an important part, each patient has to be monitored for oxygen saturation level, and this would help us analyze when a subject enters from Mild to moderate stage
Value of coagulation indicators | Day 0, Day 5±1 and Day of discharge i.e Day 10±1
  D Dimer levels has to be measured to study the D dimer levels of the patient as most researchers claiming covid-19 to be relative to coagulation. This study will help us identity the same.
Time to first negative SARS-CoV-2 PCR in NP swab | Day 0, Day 5±1 and Day of discharge i.e Day 10±1
  via ICMR recognized RT-PCR to identify when a patient is coronavirusfree
Duration of oxygen therapy | upto day 10+1
  To identify how long a patient needs oxygen therapy in certain case
Proportion of participants in each group with need for mechanical ventilation | upto day 10+1
  This is considered as a part of pharmacovigilance, as how many people enters moderate to severe case, if any
Duration of hospitalization | upto day 10+1
  most mild cases that becomes asymptomatic are sent back from hospital and treated at home quarantine. this is to identify when a patient becomes asymptomatic

CONTACTS AND LOCATIONS:
Overall Officials: Abhijit Munshi, Principal Investigator — Mittal Global Clinical Trial Services; Vijaykumar Kamat, Study Director — Corival Lifesciences Pvt Ltd; Apurve Mehra, Study Director — Biogetica
Locations (3):
- India (3):
  - Govt Medical College and Govt General Hospital (Old RIMSGGH), Srikakulam, Andhra Pradesh
  - Parul Institute of Ayurveda and Research Parul University, Vadodara, Gujarat
  - Lokmanya Hospital, Pune, Maharashtra

IPD SHARING:
Plan to Share IPD: Undecided
The trial is meant for pandemic, and any data is fruitful to the society will be shared with researchers only, without compromising personal data of the participant.

REFERENCES:
- See also: product in intervention that seeks this re-purpose study — https://immunofree.me/